CLINICAL TRIAL: NCT02184065
Title: Clinical and Therapeutic Evaluation of Meloxicam in Mexican Patients With Rheumatic Diseases
Brief Title: Observational Study of Meloxicam in Mexican Patients With Rheumatic Diseases
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 107.272
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Meloxicam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Meloxicam
  Interventions: Drug: Meloxicam

INTERVENTIONS:
Drug: Meloxicam

SUMMARY:
Observational study to evaluate the efficacy and safety of meloxicam (Mobicox®) in Mexican population with rheumatic diseases

ELIGIBILITY:
Inclusion Criteria:

* Age of 12 or older and rheumatologic disease

Exclusion Criteria:

* Hypersensitivity to meloxicam
* Hypersensitivity to other Non-steroidal anti-inflammatory drugs (NSAIDS)
* History of asthma, angioedema or urticaria secondary to NSAIDS
* Pregnancy or lactation
* Recent or current history of peptic ulcer disease, severe renal failure and severe hepatic failure

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 22639 (Actual)
Dates: Start 2004-01; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Intensity of symptoms at rest evaluated with a 4-point scale | 30 and 90 days
Intensity of symptoms during movement evaluated with a 4-point scale | 30 and 90 days
Medical global evaluation on a 4-point scale | 30 and 90 days